CLINICAL TRIAL: NCT00480116
Title: Phase III, Single Centre, Double Blind, Randomised Study Evaluating the Consistency of Three Lots of Henogen's New Adjuvanted Hepatitis B Vaccine, When Given at 0, 1 Month Schedule in Healthy Volunteers Aged 18 Years to 40 Years.
Brief Title: Consistency Study of Three Lots of Henogen's Adjuvanted Hepatitis B Vaccine When Given in 0, 1 Month Schedule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henogen (Industry)
Responsible Party: Houard, Henogen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HN016/HBV-002
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Hepatitis B
Keywords: Consistency; Immunogenicity
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Biological: Adjuvanted Hepatitis B vaccine Lot 1
- 2 (Active Comparator)
  Interventions: Biological: Adjuvanted Hepatitis B vaccine Lot 2
- 3 (Active Comparator)
  Interventions: Biological: Adjuvanted Hep B vaccine Lot 3

INTERVENTIONS:
Biological: Adjuvanted Hepatitis B vaccine Lot 1 — 20 µg, IM, month 0 and 1
  Arms: 1
Biological: Adjuvanted Hepatitis B vaccine Lot 2 — 20µg, IM, month 0 and 1
  Arms: 2
Biological: Adjuvanted Hep B vaccine Lot 3 — 20µg, IM, month 0 and 1
  Arms: 3

SUMMARY:
The study vaccine has been developed for use in pre-dialysis/ haemodialysis patients and immuno-compromised individuals who could have or had a sub-optimal response following vaccination for hepatitis B with currently available commercial vaccines (target population). This study will aim to confirm in a clinical setting the consistency of production of three lots of the vaccine.

DETAILED DESCRIPTION:
Double-blind, randomised, single centre study with three groups receiving three different lots of Henogen's adjuvanted hepatitis B vaccine according to 0, 1 months schedule. Blood samples will be taken at Month 0, Months 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female adult aged between 18 and 40 years.
* Written informed consent obtained from the subject

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Administration of a vaccine not foreseen by the study protocol within 14 days (killed vaccine) or 30 days (attenuated/ live vaccine) before the first vaccine dose.
* Concurrently participating in another clinical study or exposure to an investigational or a non-investigational product (pharmaceutical product or device).
* History of hepatitis B infection.
* Known exposure to hepatitis B virus within 6 months.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Anti-HBs seroprotection rates at Month 2. | Month 2

SECONDARY OUTCOMES:
Anti-HBs geometric mean concentration, seropositivity rates, seroprotection rates and the percentage of subjects with antibody concentrations superior or equal to 100 mIU/ml after HB-AS02V vaccination, at all time points. | Month 0, 1 and 2
Occurrence and intensity of solicited local signs and symptoms, as well as occurrence, intensity and relationship to vaccination of solicited general signs and symptoms, within 4 days after administration of study vaccine (Day 0 to 3). | Month 0 and 1
Occurrence, intensity and relationship to vaccination of unsolicited symptoms after administration of study vaccine (Day 0 to 30) | Month 0 and 1
Occurrence, intensity and relationship to vaccination of all serious adverse events (SAEs) up to Month 2. | Month 0 to 2

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Beran, MD, Principal Investigator — Vaccination and Travel Medicine Centre Poliklinika II
Locations (1):
- Vaccination and Travel Medicine Centre Poliklinika II, Hradec Králové, Czechia

REFERENCES:
- [Derived] Beran J, Hobzova L, Wertzova V, Kuriyakose S, Leyssen M, Surquin M, Houard S. Safety and immunogenicity of an investigational adjuvanted hepatitis B vaccine (HB-AS02V) in healthy adults. Hum Vaccin. 2010 Jul;6(7):578-84. doi: 10.4161/hv.6.7.11883. Epub 2010 Jul 1. PMID 20523113